CLINICAL TRIAL: NCT01061853
Title: Efficacy of Topical Rapamycin in Treatment of Chronic Erosive Oral Lichen Planus. Double Blind Randomised Controlled Trial Rapamycin vs Topical Steroids
Brief Title: Efficacy of Topical Rapamycin to Treat Chronic Erosive Oral Lichen
Acronym: RALIB
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per protocol intermediate analyses of 76 patients and enrollment difficulties.
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRN06-LV/RALIB; 2007-000152-14 (EudraCT Number)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; chronic inflammatory; mucous membranes; erosive lesions
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T (Experimental): TOPICAL SIROLIMUS AND PETROLATUM IN ORABASE
  Interventions: Drug: TOPICAL SIROLIMUS (RAPAMUNE*)
- C (Active Comparator): TOPICAL BETAMETHASONE 0.05% in ORABASE AND PHOSAL
  Interventions: Drug: TOPICAL BETAMETHASONE 0.05%

INTERVENTIONS:
Drug: TOPICAL SIROLIMUS (RAPAMUNE*) — APPLICATION ON THE LESIONS OF TOPICAL SIROLIMUS (RAPAMUNE*)1mg/ml bid during 3 months
  Arms: T
Drug: TOPICAL BETAMETHASONE 0.05% — APPLICATION ON THE LESIONS OF TOPICAL BETAMETHASONE (DIPROLENE*)0.05% bid during 3 months
  Arms: C

SUMMARY:
The purpose of this study is to determine wether topical rapamycin is more efficient than topical steroids in the treatment of chronic erosive lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* Oral Lichen Planus
* Oral Erosive Area More Than 1cm²
* Lichen Planus Pathologically Proven

Exclusion Criteria:

* No Previous Treatment by Rapamycin
* Non Child Bearing Or Breast Feeding Woman
* Patient Who Cannot Be Treated By Rapamycin Or Betamethasone
* Chronic Renal Insufficiency (Creatinin Clearance < 40ml/Mn)
* Ongoing Treatment By Topical Calcineurin Inhibitors Or Systemic Steroids Or Retinoids Or Systemic Immunosuppressors Or Thalidomide Or Griseofulvin Or Antimalarials
* Cholesterolemia >7.8 Mmol/L Or Hypertriglyceridemia >3.95mmol/L Non Responsive To Medical Treatments
* Leucopenia (<3000/Mm3)
* Thrombopenia (<100 000/Mm3)
* Hypertransaminasemia (>3n)
* Hypersensitivity To Macrolides

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
COMPLETE CLEARING OF ORAL EROSIVE LESIONS | THREE MONTHS

SECONDARY OUTCOMES:
REGRESSION OF EROSIVE SURFACE AREA | THREE MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Loïc VAILLANT, MD, Study Director — Centre 1-TOURS; Camille FRANCES, MD, Principal Investigator — Centre-2 Tenon; Scarlette AGBO-GODEAU, MD, Principal Investigator — Centre-3 La Pitié-Salpêtrière; Liliane LAROCHE, MD, Principal Investigator — Centre-4 Avicenne; Francis PASCAL, MD, Principal Investigator — Centre-5 St-Louis; Emmanuel DELAPORTE, MD, Principal Investigator — Centre-6 Lille; Alain TAÏEB, MD, Principal Investigator — Centre-7 Bordeaux; Jean-Philippe DELACOUR, MD, Principal Investigator — Centre -8 Nice; Philippe BERNARD, MD-PHD, Principal Investigator — Centre-9 REIMS
Locations (9):
- France (9):
  - University Hospital of REIMS, Reims, Marne
  - Hospital Avicenne-APHP, Bobigny
  - University Hospital of Bordeaux-St.André, Bordeaux
  - University Hospital of Lille, Lille
  - University Hospital of Nice, Nice
  - Hospital Saint Louis-APHP, Paris
  - Hospital La Pitié-Salpêtrière APHP, Paris
  - Hospital Tenon-APHP, Paris
  - University hospital of Tours, Tours